CLINICAL TRIAL: NCT07278115
Title: Effects on Remission of Type 2 Diabetes Mellitus Following Roux-en-Y Gastric Bypass Alone vs Roux-en-Y Gastric Bypass Combined With Truncal Vagotomy: A Triple-Blind Randomized Controlled Trial.
Brief Title: Effects on Remission of Type 2 Diabetes Mellitus Following Gastric Bypass Alone vs Gastric Bypass Combined With Truncal Vagotomy
Acronym: VagusSx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Research Institute for the Study of Genetic & Malignant Disorders in Childhood (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Athena Kapralou, General Surgeon, Scientific Associate, First Department of Propaedeutic Surgery, National and Kapodistrian University of Athens, University Research Institute for the Study of Genetic & Malignant Disorders in Childhood
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HippokrationHosp89/14-07-2025
Record Dates: First submitted 2025-09-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Type 2 diabetes mellitus; Insulin Resistance; Hyperglycemia; Obesity; Bariatric Surgery; Gastric Bypass; Vagotomy; Diabetes Surgery; Gut Hormones; GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Hyperglycemia; Obesity | interventions — Gastric Bypass; Vagotomy, Truncal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roux-en-Y Gastric Bypass with Truncal Vagotomy (Experimental): Participants in this arm will undergo a standard laparoscopic Roux-en-Y gastric bypass (RYGB) procedure combined with bilateral truncal vagotomy. The operation includes creation of a small gastric pouch completely separated from the remnant stomach, gastrojejunostomy to the alimentary limb, and a jejunojejunostomy to restore intestinal continuity, resulting in proximal intestinal bypass of the duodenum and proximal jejunum. Truncal vagotomy is performed by dividing both anterior and posterior vagal trunks at the lower esophagus to reduce vagally mediated biliopancreatic secretion and neurohormonal stimulation of digestion. This combined procedure aims to assess whether dual interruption of vagal and duodenal signaling enhances the metabolic and glycemic benefits of gastric bypass, promoting durable remission of type 2 diabetes mellitus.
  Interventions: Procedure: Roux-en-Y Gastric Bypass plus Truncal Vagotomy
- Roux-en-Y Gastric Bypass Alone (Active Comparator): Participants in this arm will undergo a standard laparoscopic Roux-en-Y gastric bypass (RYGB) procedure without vagotomy. The surgery includes creation of a small, completely separated gastric pouch, a gastrojejunostomy to the alimentary limb, and a jejunojejunostomy approximately 100-150 cm distal to the ligament of Treitz, resulting in a proximal intestinal bypass of the duodenum and proximal jejunum. This configuration limits nutrient exposure to the upper gut, thereby inducing metabolic changes known to improve glycemic control and weight reduction. The procedure follows established bariatric surgical principles and serves as the control arm to evaluate the additive effect of truncal vagotomy on glucose homeostasis, gut hormone secretion, and remission of type 2 diabetes mellitus.
  Interventions: Procedure: Roux-en-Y Gastric Bypass

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass plus Truncal Vagotomy — Laparoscopic Roux-en-Y gastric bypass performed according to protocol, including creation of a small gastric pouch, gastrojejunostomy, and jejunojejunostomy. In addition, bilateral truncal vagotomy is performed at the distal esophagus, dividing both anterior and posterior vagal trunks to reduce vagal stimulation of the gastrointestinal tract. The combined procedure aims to assess whether vagotomy enhances type 2 diabetes mellitus remission beyond the effect of gastric bypass alone.
  Arms: Roux-en-Y Gastric Bypass with Truncal Vagotomy
Procedure: Roux-en-Y Gastric Bypass — Laparoscopic Roux-en-Y gastric bypass performed according to protocol, including creation of a small gastric pouch, gastrojejunostomy, and jejunojejunostomy. No vagotomy is performed. This serves as the active comparator to evaluate the independent effect of adding truncal vagotomy on type 2 diabetes mellitus remission.
  Arms: Roux-en-Y Gastric Bypass Alone

SUMMARY:
This randomized, triple-blind clinical trial investigates whether adding truncal vagotomy to Roux-en-Y gastric bypass (RYGB) enhances remission of type 2 diabetes mellitus (T2DM) in patients with obesity. The study explores whether modulation of vagal signaling provides superior metabolic outcomes compared to standard RYGB alone.

Background:

RYGB is a proven metabolic procedure capable of inducing diabetes remission; however, the mechanisms remain incompletely defined. Emerging evidence supports a duodenum-centered neurohormonal model suggesting that amplified digestion-driven by vagal and hormonal hyperstimulation-plays a key role in the development of insulin resistance. The vagus nerve regulates pancreatic and biliary secretion, as well as gut hormone release. By combining truncal vagotomy with RYGB, the study aims to attenuate vagal overactivation and evaluate its impact on glucose homeostasis and hormonal adaptation.

Design:

Eligible adults (18-65 years) with BMI ≥30 kg/m² and confirmed T2DM (HbA1c ≥6.5%, or on antidiabetic therapy with HbA1c ≥6.1%) will be randomized to:

1. RYGB alone, or
2. RYGB with truncal vagotomy. Participants, postoperative staff, and assessors will remain blinded to allocation.

Primary Outcome:

Remission of T2DM at 12 months postoperatively, defined as fasting plasma glucose <100 mg/dL and HbA1c <6.0% without antidiabetic medication for at least one year.

Secondary Outcomes:

Changes in HbA1c, fasting glucose, insulin, C-peptide, OGTT-derived indices, GLP-1, CCK, PYY, GLP-2, oxyntomodulin responses, HOMA-IR, body composition, cardiovascular risk markers, medication use, and quality-of-life parameters. Surgical metrics include hospital stay, readmissions, complications, gastrointestinal symptoms, nutritional deficiencies, and bone density changes.

Follow-Up:

Assessments occur preoperatively and at 1, 3, 6, and 12 months after surgery.

Significance:

The VagusSx Trial tests whether targeted vagal and duodenal pathway interruption can improve glycemic control beyond weight loss alone, offering a novel, physiology-based strategy for durable diabetes remission.

DETAILED DESCRIPTION:
Detailed Description

This randomized, triple-blind, controlled clinical trial evaluates the metabolic impact of adding truncal vagotomy to standard Roux-en-Y gastric bypass (RYGB) in adults with obesity and type 2 diabetes mellitus (T2DM). The trial, titled VagusSx, investigates whether targeted interruption of vagal signaling augments diabetes remission beyond the effects of caloric restriction and weight loss alone.

Scientific Background and Rationale

RYGB has been established as an effective metabolic surgery leading to remission of T2DM in a significant proportion of patients. However, the exact mechanisms remain incompletely understood. Increasing evidence supports a duodenum-centered neurohormonal model in which amplified digestion-driven by chronic vagal and enteroendocrine hyperstimulation-promotes insulin resistance. The vagus nerve regulates biliopancreatic secretion, gastric motility, and the release of hormones such as cholecystokinin (CCK) and secretin. Continuous exposure to high-fat, high-glycemic diets may cause persistent vagal activation, exaggerated hormonal secretion, and enhanced nutrient absorption, ultimately contributing to β-cell stress and insulin resistance.

Truncal vagotomy is hypothesized to attenuate this hyperactivation, reducing biliopancreatic output and digestive efficiency, thereby improving glucose homeostasis and insulin sensitivity. When combined with RYGB-which excludes the duodenal mucosa from nutrient contact and enhances distal gut hormone signaling-the dual intervention may provide synergistic effects through both neural and hormonal pathways.

Study Design

This is a prospective, randomized (1:1), triple-blind clinical trial with two parallel arms:

Standard RYGB (control group)

RYGB plus truncal vagotomy (intervention group)

Participants, postoperative care staff, and assessors remain blinded to allocation. Randomization is performed via concealed envelopes using computer-generated sequences.

Eligibility

Inclusion criteria: adults aged 18-65 years, BMI ≥30 kg/m², confirmed T2DM with HbA1c ≥ 6.5% or use of antidiabetic medication with HbA1c ≥ 6.1%, and Advanced DiaRem Score > 5.

Key exclusion criteria: prior bariatric or major abdominal surgery, type 1 diabetes, chronic corticosteroid use, major psychiatric or systemic disease, or substance abuse.

Interventions

All surgeries are performed laparoscopically by the same surgical team.

Roux-en-Y gastric bypass (RYGB): creation of a small gastric pouch, gastrojejunostomy, and jejunojejunostomy (proximal intestinal bypass).

Truncal vagotomy: complete division of anterior and posterior vagal trunks at the distal esophagus prior to gastric pouch creation.

Standardized perioperative and nutritional management is applied to both groups.

Assessments and Follow-Up

Participants are evaluated at baseline (preoperative), and at 1, 3, 6, and 12 months postoperatively.

Data are collected by a multidisciplinary team (surgery, endocrinology, dietetics, psychology) using standardized laboratory, imaging, and validated questionnaires.

Primary Outcome

Remission of T2DM at 12 months, defined as fasting plasma glucose < 100 mg/dL and HbA1c < 6.0% without antidiabetic therapy for ≥12 months.

Key Secondary Outcomes

Glycemic and hormonal parameters: HbA1c, fasting glucose, insulin, C-peptide, OGTT-derived indices (insulin sensitivity, β-cell responsiveness, disposition index), and hormonal responses (GLP-1, CCK, PYY, GLP-2, oxyntomodulin).

Body composition and anthropometry: weight, BMI, waist/hip ratio, fat mass, lean mass.

Cardiometabolic risk markers: lipid profile, blood pressure, CRP, ASCVD and SCORE2-Diabetes risk indices.

Bone status: bone mineral density by DEXA.

Nutritional status: micronutrient levels (vitamins A, D, E, K, B1, B12, folate, iron, zinc, copper, calcium, magnesium, phosphorus) and prevalence of deficiencies.

Medication use: discontinuation or reduction of antidiabetic, antihypertensive, and lipid-lowering therapies.

Surgical metrics: length of stay, readmissions, early and late complications (graded by Dindo classification), gastrointestinal symptoms, dumping syndrome, and hypoglycemia episodes.

Dietary behavior: changes in food frequency, tolerance, craving, and binge-eating scales.

Physical activity: objectively measured and self-reported activity (IPAQ).

Psychosocial outcomes: treatment satisfaction, diabetes-related symptoms, and psychological well-being.

Data Management and Analysis

All data are recorded in electronic case-report forms and stored in a secure database. Continuous variables will be analyzed using repeated-measures ANOVA or mixed models. Categorical data will be compared with χ² or Fisher's exact tests. Statistical significance is set at p < 0.05. Intention-to-treat and per-protocol analyses will be performed.

Ethical Considerations

The trial adheres to the Declaration of Helsinki, Good Clinical Practice (GCP) standards, and COPE ethical guidelines. Written informed consent is obtained from all participants. The study protocol has received institutional ethics approval and is registered at ClinicalTrials.gov.

Significance

The VagusSx trial introduces a novel physiologic concept: neural-hormonal modulation of digestion as a therapeutic target in diabetes surgery. By interrupting vagal and proximal intestinal signaling, the study aims to test whether this combined intervention promotes durable diabetes remission beyond the effects of caloric restriction, potentially reshaping the mechanistic understanding and future direction of metabolic surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m²
* Age: 18-68 years
* Confirmed type 2 diabetes mellitus with:

  * HbA1c ≥ 6.5%, or
  * HbA1c ≥ 6.1% and the use of antidiabetic medication
* Advanced-DiaRem Score > 5* * Advanced-DiaRem Score: a validated scoring system predicting diabetes remission after bariatric surgery.

Exclusion Criteria:

* Previous bariatric surgery or major abdominal surgery (e.g., enterectomy, gastrectomy, colectomy, hepatectomy, partial or total pancreatectomy)
* Major, uncompensated health problems (major psychiatric, endocrine, cardiac, pulmonary, hepatic, or renal disorder; cancer; or other conditions with increased risk of complications)
* Use of corticosteroids (glucocorticoids):

  * Chronic corticosteroid use for > 3 months within the last year, or
  * Corticosteroid therapy within the last 3 months
* Type 1 diabetes mellitus
* Alcohol or drug addiction

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Complete remission of Type 2 Diabetes Mellitus at 12 Months Post-Surgery | 12 months postoperatively
  Complete remission of type 2 diabetes will be defined as fasting plasma glucose <100 mg/dL and HbA1c <6.0%, maintained without the use of any antidiabetic medications for at least one year following surgery.

SECONDARY OUTCOMES:
Partial remission of type 2 diabetes | 12 months postoperatively
  Partial remission will be defined as HbA1c < 6.5% and fasting plasma glucose between 100-125 mg/dL, maintained without the use of any antidiabetic medications for at least one year following surgery.
Fasting Plasma Glucose | Baseline and up to 12 months postoperatively
  Change in fasting plasma glucose levels will be measured at each follow-up visit (1, 3, 6, and 12 months).
Fasting Insulin | Baseline and 12 months postoperatively
  Change in fasting insulin levels will be assessed at baseline (pre-surgery) and at 12 months after surgery.
Fasting C-Peptide levels | Baseline and 12 months postoperatively
  Change in fasting C-peptide levels will be assessed at baseline (pre-surgery) and at 12 months postoperatively.
HbA1c | Baseline, 1, 3, 6, and 12 months postoperatively
  Change in HbA1c (%) from baseline across follow-up visits.
Oral Glucose Tolerance Test (OGTT) Indices-plasma glucose measurement | Baseline and 12 months postoperatively
  After an overnight fast, participants will ingest 75 g of glucose orally. Blood samples will be collected at baseline (fasting) and at regular time intervals over a two-hour period, post-pradially to measure plasma glucose, insulin, and C-peptide.
HOMA-IR (Insulin Resistance Index) | Baseline and 12 months postoperatively
  The Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) will be calculated using fasting plasma glucose and fasting insulin levels, according to the following formula:
  HOMA-IR=Fasting glucose (mg/dL)×0.0555×Fasting insulin (mU/L)/22.5
Use of Antidiabetic Medications | Baseline, 1, 3, 6, and 12 months postoperatively
  Change in the number of antidiabetic medications prescribed per patient compared with baseline. Each active oral or injectable non-insulin agent will be counted as one medication. A decrease in the number of medications will be considered an indicator of improved glycemic control.
  Unit of Measure: Number of medications per participant
Use of Insulin Therapy | Baseline, 1, 3, 6, and 12 months postoperatively
  Change in insulin therapy status at each follow-up visit, expressed as the proportion of participants achieving:
  Complete discontinuation of insulin therapy,
  ≥50% reduction in daily insulin dose, or No change / continued insulin requirement. The primary reported measure will be the percentage of participants discontinuing insulin therapy, with additional categorical data on dose reduction and continuation summarized descriptively.
  Unit of Measure:
  Percentage of participants (%)
Body Weight | Baseline, 1, 3, 6, and 12 months postoperatively
  Change in body weight (kg) from baseline at each follow-up visit, measured under standardized conditions.
Body Mass Index (BMI) | Baseline, 1, 3, 6, and 12 months postoperatively
  Change in BMI (kg/m²) calculated from measured weight and height at each visit.
Waist and Hip Circumference | Baseline, 1, 3, 6, and 12 months postoperatively
  Change in waist and hip circumference (cm) measured with a flexible tape at standardized anatomical landmarks; waist-to-hip ratio will also be derived.
Body Composition | Baseline and 12 months postoperatively
  Change in body fat percentage (% body fat) from baseline to 12 months postoperatively.
Total Cholesterol | Baseline, 1, 3, 6, and 12 months postoperatively
  Change in fasting total cholesterol (mg/dL) measured by standard enzymatic methods.
HDL Cholesterol | Baseline, 1, 3, 6, and 12 months postoperatively
  Change in fasting high-density lipoprotein cholesterol (mg/dL).
LDL Cholesterol | Baseline, 1, 3, 6, and 12 months postoperatively
  Change in fasting low-density lipoprotein cholesterol (mg/dL).
Triglycerides | Baseline, 1, 3, 6, and 12 months postoperatively
  Change in fasting triglyceride levels (mg/dL).
C-Reactive Protein (CRP) | Baseline, 1, 3, 6, and 12 months postoperatively
  Change in high-sensitivity C-reactive protein (mg/L) as a marker of systemic inflammation.
Blood Pressure | Baseline, 1, 3, 6, and 12 months postoperatively
  Change in systolic and diastolic blood pressure (mmHg).
Change in Use of Lipid-Lowering Medications | Baseline, 1, 3, 6, and 12 months postoperatively
  Change in the proportion of participants using lipid-lowering medications compared to baseline. Medication use status (continued, reduced dose, or discontinued) will be assessed at each postoperative visit.
Use of Antihypertensive Medications | Baseline, 1, 3, 6, and 12 months postoperatively.
  Change in the number and classes of antihypertensive drugs prescribed.
Cardiovascular Risk Index (Obesity-Related) | Baseline and 12 months postoperatively
  Change in obesity-related cardiovascular risk, assessed using the ASCVD (Atherosclerotic Cardiovascular Disease) Risk Score developed by the American College of Cardiology. Calculation will be performed using the official online tool: https://tools.acc.org/ascvd-risk-estimator-plus/#!/calculate/estimate/.
Cardiovascular Risk Index (Diabetes-Related) | Baseline and 12 months postoperatively
  Change in cardiovascular risk related to diabetes, assessed using the SCORE2-Diabetes risk prediction model, developed, calibrated, and validated by the European Society of Cardiology (ESC). Calculation will be performed through the ESC online tool: https://www.escardio.org/Education/ESC-Prevention-of-CVD-Programme/Risk-assessment/esc-cvd-risk-calculation-app.
Oral Glucose Tolerance Test (OGTT) Indices-plasma insulin measurement | Baseline and 12 months postoperatively
  After an overnight fast, participants will ingest 75 g of glucose orally. Blood samples will be collected at baseline (fasting) and at regular time intervals over a two-hour period, post-pradially to measure plasma insulin.
Oral Glucose Tolerance Test (OGTT) Indices-plasma C-peptide levels | Baseline and 12 months postoperatively
  After an overnight fast, participants will ingest 75 g of glucose orally. Blood samples will be collected at baseline (fasting) and at regular time intervals over a two-hour period, post-pradially to measure plasma C-peptide.
Discontinuation of Antidiabetic Medications | Baseline, 1, 3, 6, and 12 months postoperatively
  Proportion of participants who discontinue all antidiabetic medications (excluding insulin) following surgery while maintaining normoglycemia.
  Unit of Measure: Percentage of participants (%)

OTHER OUTCOMES:
Postprandial Hormonal and Glucose Response to Mixed-Meal Test | Baseline and 12 months postoperatively
  After a 12-hour overnight fast, participants will undergo a standardized mixed-meal test. The test meal (800 kcal total) consists of a solid portion (one egg, two slices of white bread, and 5 g margarine; ~250 kcal) and a liquid portion (200 mL cream with 2 teaspoons chocolate powder; ~550 kcal), consumed within 5 minutes. Blood samples will be collected at baseline (fasting) and at regular time intervals over a three-hour period, post-pradially. Plasma concentrations of glucose, insulin, cholecystokinin (CCK), glucagon-like peptide-1 (GLP-1), peptide YY (PYY), glucagon-like peptide-2 (GLP-2), and oxyntomodulin will be measured to evaluate the postprandial metabolic and hormonal response.
Prevalence of Micronutrient Deficiencies | Baseline, 1, 3, 6, and 12 months postoperatively (selected micronutrients per protocol schedule)
  Proportion of participants presenting with one or more micronutrient deficiencies. Deficiencies will be defined according to standard laboratory reference ranges for each micronutrient (e.g., vitamin B12, folate, vitamin D, iron, ferritin, zinc, copper, vitamins A, E).
  Blood samples will be obtained per protocol at baseline and follow-up visits (specific micronutrients assessed at 3, 6, or 12 months, as indicated)
Obstructive Sleep Apnea Score | Baseline and 12 months postoperatively
  Change in obstructive sleep apnea risk assessed using the STOP-Bang questionnaire (http://www.stopbang.ca/osa/screening.php).
Early Postoperative Complications | Up to 6 weeks postoperatively
  Evaluation of early postoperative surgical complications graded according to the Clavien-Dindo classification.
Late Postoperative Complications | Beyond 6 weeks postoperatively
  Evaluation of late postoperative surgical complications, graded according to the Clavien-Dindo classification.
Length of Hospital Stay | Index hospitalization (from day of surgery until discharge)
  Duration of initial postoperative hospitalization, expressed in calendar days from the date of surgery (Day 0) to the date of discharge. Both mean and median length of stay, along with interquartile ranges, will be reported.
  Prolonged hospitalizations related to postoperative complications will also be recorded and analyzed separately.
  Unit of Measure:
  Days
Unplanned Hospital Readmissions | Within 30 days and up to 12 months postoperatively
  Incidence of unplanned hospital readmissions related to the index surgical procedure. Readmissions are defined as any unscheduled overnight hospital stay following discharge, excluding planned follow-up or elective admissions. Both early (≤30 days) and late (>30 days to 12 months) readmissions will be recorded, with cause and timing documented.
Surgery-Related Events | From the day of surgery up to 12 months postoperatively
  Recording and classification of any surgical events directly or indirectly related to the operative procedure. This includes intraoperative events (e.g., bleeding, injury to adjacent organs), early postoperative events (e.g., anastomotic leak, wound infection), and late complications (e.g., stricture, internal hernia). Events will be documented and categorized according to their timing and clinical relevance.
Medical Events Related to Surgery | From the day of surgery up to 12 months postoperatively
  Recording of medical conditions that arise directly or indirectly in association with the surgical intervention. This includes events such as pulmonary complications (e.g., pneumonia, atelectasis), thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism), cardiovascular complications (e.g., arrhythmias, myocardial infarction), or metabolic disturbances (e.g., electrolyte imbalances, malnutrition). All events will be documented, classified, and analyzed in relation to their potential link to the surgical procedure.
Diabetes-Related Complications | From the day of surgery up to 12 months postoperatively
  Occurrence of acute and chronic complications directly associated with type 2 diabetes mellitus. This includes hypoglycemic episodes, diabetic ketoacidosis, hyperosmolar states, infections with impaired wound healing, and progression or new onset of microvascular (retinopathy, nephropathy, neuropathy) or macrovascular complications. All events will be systematically recorded, graded, and analyzed in relation to the postoperative course.
Hypoglycemia Episodes | From baseline through 12 months postoperatively
  ypoglycemia will be assessed based on patient-reported symptoms, using the 11 most frequent clinical manifestations described in the Edinburgh Hypoglycemia Scale. These include: Autonomic Nervous System Symptoms: sweating, palpitations, tremor, hunger Neuroglycopenic Symptoms: confusion, drowsiness, abnormal behavior, speech difficulty, incoherence General Malaise: headache, nausea Episodes will be systematically captured and evaluated with the modified Clarke Hypoglycemia Questionnaire, adapted for patients with type 2 diabetes mellitus. The scoring range is 2-46 points, with higher scores reflecting greater hypoglycemia risk and severity.
Dumping Syndrome Assessment | Baseline, 1, 3, 6, and 12 months postoperatively
  The presence and severity of dumping syndrome will be evaluated using two validated scoring systems:
  Sigstad's Score - Traditionally applied in peptic ulcer surgery, bariatric surgery, and upper gastrointestinal surgery. It is primarily used for the identification of early dumping syndrome.
  Arts Dumping Score Questionnaire - Used to differentiate early from late dumping syndrome and to quantify the severity of symptoms.
  These tools will enable systematic identification of clinically significant dumping symptoms and monitoring of their progression over time.
Gastrointestinal Symptoms | Baseline, 1, 3, 6, and 12 months postoperatively
  Gastrointestinal symptoms will be assessed using the Gastrointestinal Symptom Rating Scale (GSRS), as adapted for gastric bypass patients. This validated questionnaire evaluates the frequency and severity of common gastrointestinal complaints, providing a standardized measure of postoperative changes in digestive function.
Screening for Micronutrient Deficiencies | Baseline, 3, 6, and 12 months postoperatively (frequency depending on the nutrient, per ASMBS guidelines and the study protocol
  Patients will undergo systematic preoperative and postoperative screening of vitamin and mineral levels in order to identify and correct deficiencies, in accordance with the American Society for Metabolic and Bariatric Surgery (ASMBS) guidelines. This includes assessment of key micronutrients such as fat- and water-soluble vitamins (A, D, E, K, B12, folate), iron, calcium, magnesium, zinc, and phosphorus.
Bone Mineral Density | Baseline and 12 months postoperatively
  Bone mineral density will be assessed using dual-energy X-ray absorptiometry (DEXA). The outcome will evaluate changes in bone density to monitor potential skeletal effects of surgery.
Meal Frequency and Food Intake Patterns (Food Frequency Questionnaire - FFQ) | Baseline and 12 months postoperatively
  Change in dietary intake patterns assessed using the Food Frequency Questionnaire (FFQ). The FFQ evaluates the frequency, type, and portion of foods consumed to identify shifts in caloric intake, macronutrient composition, and eating habits following surgery.
  Unit of Measure: FFQ score (frequency scale)
Self-Reported Physical Activity | Baseline and 12 months postoperatively
  Self-reported physical activity will be assessed using the short version of the International Physical Activity Questionnaire (IPAQ-short form).
Diabetes Treatment Satisfaction | Baseline and 12 months postoperatively
  Treatment satisfaction will be assessed using the Diabetes Treatment Satisfaction Questionnaire (DTSQ). The instrument includes 8 items that measure patients' overall satisfaction with their diabetes therapy, perceived convenience, understanding of treatment, and willingness to continue. For the purposes of this study, the questionnaire has been adapted to reflect surgical treatment of diabetes rather than pharmacological management.
Diabetes-Related Symptoms | Baseline and 12 months postoperatively
  The Type 2 Diabetes Symptom Checklist (DSC-T2) will be used to evaluate the severity and frequency of diabetes-related symptoms.
Psychological Distress | Baseline and 12 months postoperatively.
  Psychological distress and depressive symptoms will be assessed using the Beck Depression Inventory-II (BDI-II).
Food Tolerance (Food Tolerance Questionnaire - FTQ) | Baseline and 12 months postoperatively
  Change in food tolerance and gastrointestinal comfort assessed by the Food Tolerance Questionnaire (FTQ). Participants rate their ability to tolerate different food textures and types (e.g., meats, dairy, fibrous foods) after surgery.
  Unit of Measure: FTQ total score.
Food Craving and Motivation (Food Craving Questionnaire - FCQ) | Baseline and 12 months postoperatively
  Assessment of craving intensity and motivational drive toward specific foods using the Food Craving Questionnaire (FCQ). The FCQ evaluates both the frequency and emotional triggers associated with cravings after metabolic surgery.
  Unit of Measure: FCQ total score
Binge Eating Behavior (Binge Eating Scale - BES) | Baseline and 12 months postoperatively
  Evaluation of binge eating behavior using the Binge Eating Scale (BES). The BES assesses the presence and severity of binge eating episodes and emotional eating patterns, with higher scores indicating more severe binge behavior.
  Unit of Measure: BES score (points)

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Surgery, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Yes. Individual participant data (IPD) that underlie the results reported in future publications will be shared, including de-identified datasets of baseline characteristics, perioperative data, and postoperative outcomes (glycemic indices, weight, laboratory results, complications, and follow-up measures). A data dictionary describing all variables will also be provided to allow full interpretation. Data will be available to qualified researchers upon reasonable request and with approval from the coordinating center at Hippokration University Hospital.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months after publication of the primary results with no end date.
Access Criteria: De-identified individual participant data (IPD) and supporting documents (Study Protocol, Statistical Analysis Plan, Informed Consent Form) will be available to qualified researchers affiliated with Hippokration University Hospital. Access will be granted for scientifically valid analyses that are consistent with the objectives of the VagusSx trial, particularly in the fields of diabetes, obesity, metabolic surgery, and related endocrine or cardiovascular outcomes.
  Requests must include a research proposal outlining study objectives, statistical methods, and a data management plan. All requests will be reviewed by the VagusSx Trial Steering Committee at Hippokration University Hospital to ensure scientific merit, ethical compliance, and alignment with participant consent.
  Approved researchers will be required to sign a data sharing agreement to protect confidentiality and limit use of the data to the approved project. Data will be provided in ele

REFERENCES:
- [Background] Kapralou AN, Yapijakis C, Chrousos GP. The Duodenum-Centered Neurohormonal Hypothesis of Type 2 Diabetes: A Mechanistic Review and Therapeutic Perspective. Curr Issues Mol Biol. 2025 Aug 14;47(8):657. doi: 10.3390/cimb47080657. PMID 40864811
- [Background] Kapralou AN, Chrousos GP. Metabolic effects of truncal vagotomy when combined with bariatric-metabolic surgery. Metabolism. 2022 Oct;135:155263. doi: 10.1016/j.metabol.2022.155263. Epub 2022 Jul 11. PMID 35835160
- See also: Detailed information about the VagusSx Clinical Trial evaluating the effects of Roux-en-Y Gastric Bypass with or without Truncal Vagotomy on remission of Type 2 Diabetes Mellitus in patients with obesity. — https://diabetes.surgery/clinical-trial-vagus-sx
- See also: Peer-reviewed article by our research team (who also registered this clinical trial) exploring the metabolic effects of truncal vagotomy when combined with gastric bypass, providing mechanistic support for this novel surgical strategy in type 2 diabetes. — https://pubmed.ncbi.nlm.nih.gov/35835160/
- See also: Official website of the A' Department of Propaedeutic Surgery, School of Medicine, National and Kapodistrian University of Athens, based at Hippocration General Hospital of Athens - the site where the clinical trial will be conducted. — https://aproposurg.med.uoa.gr/